CLINICAL TRIAL: NCT06149637
Title: Comparison of Two Routes of Surgical Approach to Lateral Cervical Node Dissection in Differentiated Thyroid Cancer Patients With Lateral Metastatic Disease: Randomized Clinical Trial
Brief Title: Lateral Cervical Node Dissection in Differentiated Thyroid Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Excelencia en Enfermedades de Cabeza y Cuello (Other)
Collaborators: Hospital Alma Mater de Antioquia (Unknown); Hospital San Vicente Fundación (Other); Clinica Las Vegas- Grupo QuironSalud (Unknown)
Responsible Party: Principal Investigator, Alvaro Sanabria, Primary Researcher, Centro de Excelencia en Enfermedades de Cabeza y Cuello
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IN53-2021
Record Dates: First submitted 2023-08-06; First posted 2023-11-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Cancer
Keywords: neck dissection; shoulder disfunction; randomized clinical trial
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, multicenter stratified clinical trial with 1:1 allocation.
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional neck dissection approach (Active Comparator): Traditional neck dissection approach
  Interventions: Procedure: Traditional neck dissection approach
- Anterior neck dissection approach (Experimental): Anterior neck dissection
  Interventions: Procedure: Anterior neck dissection approach

INTERVENTIONS:
Procedure: Traditional neck dissection approach — .1. A transverse cervical incision is made with horizontal extension towards the affected side. 2. It is dissected through the subplatysmal plane, the posterior edge of the sternocleidomastoid muscle is dissected along its entire length. 3. Identification and dissection of the spinal nerve at Erb's point. 4. Level V nodes are dissected up to the spinal nerve without identifying or dissecting it 5. The jugular chain nodes are identified and the left level IV nodes are dissected with special attention to ligate the lymphatics of this level 6. Identification and dissection of level III nodes 7. Identification and dissection of level IIA and IIB ganglia with identification and preservation of the accessory nerve.
  Arms: Traditional neck dissection approach
Procedure: Anterior neck dissection approach — 1. A transverse cervical incision is made with horizontal extension towards the affected side.
  2. It is dissected through the subplatysmal plane, the anterior edge of the sternocleidomastoid muscle is dissected along its entire length.
  3. Level V nodes are dissected up to the spinal nerve without identifying or dissecting it
  4. The jugular chain nodes are identified and the left level IV nodes are dissected with special attention to ligate the lymphatics of this level
  5. Identification and dissection of level III nodes
  6. Identification and dissection of level IIA and IIB nodes with identification and preservation of the accessory nerve.
  Arms: Anterior neck dissection approach

SUMMARY:
The objective of this study is to compare shoulder and neck morbidity and the effectiveness of cervical lateral nodal dissection in patients with differentiated thyroid cancer and lateral metastases between the anterior and posterior approaches to the sternocleidomastoid muscle (SCM)

DETAILED DESCRIPTION:
The incidence of thyroid cancer has increased in recent decades, being responsible for 586,000 cases worldwide, ranking ninth in incidence in 2020. The rapid increase of thyroid cancer, particularly papillary thyroid cancer, has been largely attributed to the increasing use of ultrasound, along with increased use of other imaging modalities.

Similarly, analyzing the pattern of lymph node dissemination of well-differentiated thyroid carcinoma, Eskander et al., 2 reviewed all the pertinent literature up to 2011 (a total of 1,145 patients and 1,298 neck dissections) and reported an overall metastasis rate in patients taken to to surgery of 53.1%, 15.5%, 70.5%, 66.3%, 7.9% and 21.5% in levels IIa, IIb, III, IV, Va and Vb, respectively. For the Thus, the primary surgical treatment for lateral neck disease generally includes lateral neck dissection in conjunction with total thyroidectomy. Lymph node dissection should be performed in patients with biopsy-proven metastatic lateral cervical nodes. Jugular nodes located at levels II, III, and IV are the lateral neck compartments most commonly affected by CBDT and should be included in all therapeutic lateral neck dissections. Level V, which represents the posterior triangle of the neck, is affected less frequently. However, the Vb level must be dissected along with the other levels, and careful visualization and dissection of the spinal accessory nerve is paramount. Level V can be approached by an anterior approach by retracting the sternocleidomastoid muscle posteriorly, or by dissecting the posterior triangle behind the muscle sternocleidomastoid to the trapezius muscle. The precise extent of the neck dissection is a decision made based on the volume and location of the disease. The ATA recommends complete lymph node dissection (CLND), including levels II and V, for most patients with clinically evident lateral neck metastatic disease, although nuances regarding the extent of level V dissection are not clarified, in relation to whether level V should be included. Regarding the difference between the surgical techniques, the posterior approach to the sternocleidomastoid muscle involves a longer incision, where the dissection proceeds from the anterior edge of the trapezius muscle in a medial direction that includes the lymphatic contents of the supraclavicular fossa. The upper margin of this area presents the greatest risk of damage to the spinal accessory nerve. Furthermore, during the dissection of this region, several supraclavicular branches of the cervical plexus can be found. Some branches of the deep cervical plexus follow a course similar to that of the accessory nerve and may confuse the novice surgeon. In the case of the anterior approach, the incision is made up to the anterior edge of the ECM and once the accessory nerve has been identified at its insertion in the sternocleidomastoid, its course is traced superiorly to the posterior belly of the digastric. However, the effect of the anterior approach on the lymph node count and the risk of future recurrence at level V is uncertain. With these differences in terms of the approach in these two techniques, a greater length of skin incision, and greater dissection of the accessory nerve can be observed. and of the deep cervical plexus given the similar course to the XI nerve in the posterior approach, the question arises as to whether the surgical approach influences the patient's morbidity.

The main objective of the present study was to compare the morbidity and effectiveness measured in terms of lymph node count of emptying levels II to V by the anterior versus the posterior route in patients with well-differentiated thyroid cancer with lateral metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years.
2. Patients with macroscopic lymph node involvement identified by physical examination, imaging or intraoperatively in lateral neck.
3. Patients with microscopic nodal involvement confirmed by FNAB (definition by the pathologist of suspected or confirmed metastatic papillary carcinoma according to the Bethesda criteria)
4. Candidates for lateral lymph node dissection due to suspected or confirmed disease metastatic lymph nodes as defined by the treating surgeon.
5. Patients requiring or not requiring thyroidectomy and/or central dissection concomitant with the dissection

Exclusion Criteria:

1. Patients with a history of previous neck dissection
2. Histological confirmation of medullary or anaplastic carcinoma
3. Previous spinal nerve injury

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder dysfunction | 2 weeks, 3 months, 6 months, and 1 year
  (SPADI shoulder pain and disability questionnaire, validated in Spanish) Minimun score 0, maximun 100, a higher score means higher disability
Cervical disconfort | 2 weeks, 3 months, 6 months, and 1 year
  The Cervical Disability Index (IDC) validated in Spanish Minimun score 0, maximun 50, a higher score means higher disability
Complications | 30 days
  Temporary or permanent accessory nerve injury measured in the physical examination by limitation of the lateral range of movement of the shoulder less than 50%
  * Bleeding defined by the treating surgeon by physical examination
  * Wound infection: infection in the first 30 days after surgery, diagnosed with at least one of the following criteria: presence of purulent discharge from the surgical wound, presence of microorganisms isolated by taking a culture of wound discharge , presence of at least one of the signs and symptoms of inflammation (pain, redness, edema, heat).
  * Chylous fistula defined as milky discharge from the cervical drain with a triglyceride count higher than the serum.
  * Mortality
  * Re Operation before 30 days

SECONDARY OUTCOMES:
Total lymph node count. | 30 days
  Total number of resected and compromised lymph nodes according to the histopathology report
Surgical time | 30 days
  Surgical time in minutes according to the surgical report
Lateral lymph node recurrence | 5 years
  Number of participants with presence of tumor in the neck lymph nodes detected during follow-up by physical examination or imaging 6 months or more after primary surgery and confirmed cytopathologically.
Dynamic response | 5 years
  Number of participants with excellent, incomplete biochemical, incomplete structural or undetermined response according to the ATA classification.
Overall and disease-free survival | 5 years
  Overall and disease-free survival measured from the day of surgery until recurrence or termination of follow-up.
Length of postoperative hospital stay. | 30 days
  Length of postoperative hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Sanabria, Principal Investigator — Universidad de Antioquia
Locations (1):
- Hospital Alma Mater de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No